CLINICAL TRIAL: NCT01406249
Title: A Randomized Phase II Trial Comparing Capecitabine/CDDP(XP) and S-1/CDDP(SP) as the First-line Treatment for Advanced Gastric Cancer (XParTS II)
Brief Title: XParTS II: Capecitabine/CDDP(XP) and S-1/CDDP(SP) as the First-line Treatment for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECRIN-GC1107-XParTS II; UMIN000006045 (Other: UMIN Clinical Trials Registry)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer
Keywords: unresectable gastric cancer; recurrent gastric cancer; StageIV gastric cancer; adenocarcinoma of the stomach; XP; SP
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-1,Cisplatin (Active Comparator)
  Interventions: Drug: SP
- Capecitabine, Cisplatin (Experimental)
  Interventions: Drug: XP

INTERVENTIONS:
Drug: SP — Drug: S-1:
  S-1 will be administered at 40 mg/m2 orally, twice daily (80 mg/m2 total daily dose) on Days 1 through 21 of each 35-day treatment cycle.
  Drug: Cisplatin:
  Cisplatin will be administered at 60 mg/m2 by intravenous infusion on Day 8 of each 35-day treatment cycle.
  Arms: S-1,Cisplatin
Drug: XP — Drug: Capecitabine:
  Capecitabine will be administered at 1,000 mg/m2 orally, twice daily (2,000 mg/m2 total daily dose) on Days 1 through 14 of each 21-day treatment cycle.
  Drug: Cisplatin:
  Cisplatin will be administered at 80 mg/m2 by intravenous infusion on Day 1 of each 21-day treatment cycle.
  Arms: Capecitabine, Cisplatin

SUMMARY:
The aim of this study is to elucidate the efficacy and safety of XP and SP for first-line treatment of Advanced Gastric Cancer.

DETAILED DESCRIPTION:
XP and SP are either standard treatment for advanced gastric cancer. The aim of this study is to elucidate the efficacy and safety of Capecitabine/Cisplatin and S-1/Cisplatin for first-line treatment of Advanced Gastric Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma with unresectable metastatic or recurrent disease
2. Lesions confirmed on imaging within 28 days before registration (not required measurable lesions as defined in RECIST version 1.1)
3. No previous chemotherapy or radiotherapy. However, adjuvant chemotherapy is allowed the case of more than 6 months from the end of adjuvant chemotherapy
4. ECOG Performance Status of 0 to 2
5. Life expectancy of at least 3 months after registration
6. Written informed consent
7. Age of 20 to 74 years with either gender
8. Adequate Major organ functions within 14 days before registration

Exclusion Criteria:

1. Positive HER2 status
2. Previous history of fluoropyrimidines therapy within 6 months prior to registration
3. Previous treatment with platinum agents
4. Previous history of serious hypersensitivity to fluoropyrimidines or platinum agents
5. Previous history of adverse reactions suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency
6. More than one cancer at the same time or more than one cancer at different times separated by a 5-year disease-free interval. However, multiple active cancers do not include carcinoma in situ or skin cancer which is determined to have been cured as a result of treatment.
7. Obvious infection or inflammation (pyrexia ≥ 38.0˚C)
8. Active hepatitis
9. Heart disease that is serious or requires hospitalization, or history of such disease within past year
10. Having complication that is serious or requires hospitalization (intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, poorly controlled diabetes mellitus, renal failure, liver disorders, or hepatic cirrhosis)
11. Being treated or in need of treatment with flucytosine, phenytoin or warfarin potassium
12. Chronic diarrhea (watery stool or ≥4 times/day)
13. Active gastrointestinal bleeding
14. Body cavity fluids requiring drainage or other treatment
15. Clinical suspicion or previous history of metastasis to brain or meninges
16. Women who are pregnant, breastfeeding, or potentially (hoping to become) pregnant
17. Unwillingness to practice contraception
18. Poor oral intake
19. Psychiatric disorders which are being or may need to be treated with psychotropics
20. Otherwise determined by investigators or site principal investigators to be unsuitable for participation in study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | at 24weeks from patient enrollment

SECONDARY OUTCOMES:
Time-to treatment failure | 3year
Response rate | 3 year
Overall survival | 3 year
Safety | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Akira Tsuburaya, Principal Investigator — Shonan Kamakura Hospital
Locations (1):
- Epidemiological and Clinical Research Information Network, Kyoto, Japan

REFERENCES:
- [Derived] Tsuburaya A, Morita S, Kodera Y, Kobayashi M, Shitara K, Yamaguchi K, Yoshikawa T, Yoshida K, Yoshino S, Sakamoto J. A randomized phase II trial to elucidate the efficacy of capecitabine plus cisplatin (XP) and S-1 plus cisplatin (SP) as a first-line treatment for advanced gastric cancer: XP ascertainment vs. SP randomized PII trial (XParTS II). BMC Cancer. 2012 Jul 23;12:307. doi: 10.1186/1471-2407-12-307. PMID 22824079